CLINICAL TRIAL: NCT03248440
Title: A Multi-Center, Double-Masked, Randomized, Placebo-Controlled Evaluation of the Safety and Efficacy of SUN-131 Transdermal System (TDS) as Compared to Placebo TDS in Patients With a Chalazion (SUN-131-03)
Brief Title: Safety and Efficacy Study of SUN-131 Transdermal System (TDS) as Compared to Placebo TDS in Patients With a Chalazion
Acronym: SUNRISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Senju USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUN-131-03
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Chalazion
MeSH Terms: conditions — Chalazion | interventions — tyramine-deoxysorbitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SUN-131 1.5% TDS (Experimental)
  Interventions: Drug: SUN-131 1.5% TDS
- Placebo TDS (Placebo Comparator)
  Interventions: Drug: Placebo TDS

INTERVENTIONS:
Drug: SUN-131 1.5% TDS — SUN-131 1.5% TDS will be worn for 14 days
  Arms: SUN-131 1.5% TDS
Drug: Placebo TDS — No active substance; Placebo TDS will be worn each day for 14 days
  Arms: Placebo TDS

SUMMARY:
This protocol for SUN-131 1.5% TDS is developed for the treatment of chalazion. SUN-131 1.5% TDS is designed for local delivery of a corticosteroid, to the upper or lower eyelid. The purpose of this study is to evaluate the efficacy and safety of SUN-131 1.5% TDS as compared with placebo TDS in the treatment of a chalazion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 6 years of either sex and of any race
2. Subjects with a diagnosis of a single chalazion
3. Subjects with chalazion erythema score of ≥ 1
4. Normal eyelid function without active signs of eye and eyelid infection in either eye.
5. Must be willing and able to correctly apply and wear a transdermal patch to the eyelid
6. Avoid wearing contact lenses in the study eye

Exclusion Criteria:

1. Chalazion that has atypical features (a recurring chalazion at the same spot, abnormal surrounding lid tissue, associated loss of tissues).
2. History of chalazion incision and curettage in study eyelid.
3. Multiple chalazia in any one eyelid.
4. Active ocular or eyelid infection Presence of hordeolum in any one eyelid.
5. An abnormal skin condition on the study eyelid region (e.g., eczema, psoriasis, atopic dermatitis, etc.) where the study drug will be applied.
6. Diagnosed with glaucoma in either eye.
7. History of steroid-induced elevation of IOP.
8. Female subjects who are pregnant or lactating.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (59):
  - SUN-131-03 Investigational Site, Chandler, Arizona
  - SUN-131-03 Investigational Site, Prescott, Arizona
  - SUN-131-03 Investigational Site, Sun City, Arizona
  - SUN-131-03 Investigational Site, Glendale, California
  - SUN-131-03 Investigational Site, Lancaster, California
  - SUN-131-03 Investigational Site, Long Beach, California
  - SUN-131-03 Investigational Site, Los Angeles, California
  - SUN-131-03 Investigational Site, Mission Hills, California
  - SUN-131-03 Investigational Site, Petaluma, California
  - SUN-131-03 Investigational Site, Rancho Cordova, California
  - SUN-131-03 Investigational Site, San Diego, California
  - SUN-131-03 Investigational Site, Santa Ana, California
  - SUN-131-03 Investigational Site, Colorado Springs, Colorado
  - SUN-131-03 Investigational Site, Littleton, Colorado
  - SUN-131-03 Investigational Site, Fort Myers, Florida
  - SUN-131-03 Investigational Site, Largo, Florida
  - SUN-131-03 Investigational Site, Maitland, Florida
  - SUN-131-03 Investigational Site, Tamarac, Florida
  - SUN-131-03 Investigational Site, Albany, Georgia
  - SUN-131-03 Investigational Site, Morrow, Georgia
  - SUN-131-03 Investigational Site, Roswell, Georgia
  - SUN-131-03 Investigational Site, Chicago Ridge, Illinois
  - SUN-131-03 Investigational Site, Glenview, Illinois
  - SUN-131-03 Investigational Site, Hoffman Estates, Illinois
  - SUN-131-03 Investigational Site, Lake Villa, Illinois
  - SUN-131-03 Investigational Site, Leawood, Kansas
  - SUN-131-03 Investigational Site, Shawnee Mission, Kansas
  - SUN-131-03 Investigational Site, Lexington, Kentucky
  - SUN-131-03 Investigational Site, Louisville, Kentucky
  - SUN-131-03 Investigational Site, Saint Joseph, Michigan
  - SUN-131-03 Investigational Site, Bloomington, Minnesota
  - SUN-131-03 Investigational Site, Kansas City, Missouri
  - SUN-131-03 Investigational Site, St Louis, Missouri
  - SUN-131-03 Investigational Site, Washington, Missouri
  - SUN-131-03 Investigational Site, Las Vegas, Nevada
  - SUN-131-03 Investigational Site, Wantagh, New York
  - SUN-131-03 Investigational Site, Asheville, North Carolina
  - SUN-131-03 Investigational Site, Charlotte, North Carolina
  - SUN-131-03 Investigational Site, High Point, North Carolina
  - SUN-131-03 Investigational Site, Cincinnati, Ohio
  - SUN-131-03 Investigational Site, Mason, Ohio
  - SUN-131-03 Investigational Site, Lancaster, Pennsylvania
  - SUN-131-03 Investigational Site, Philadelphia, Pennsylvania
  - SUN-131-03 Investigational Site, Wayne, Pennsylvania
  - SUN-131-03 Investigational Site, Florence, South Carolina
  - SUN-131-03 Investigational Site, Rapid City, South Dakota
  - SUN-131-03 Investigational Site, Chattanooga, Tennessee
  - SUN-131-03 Investigational Site, Memphis, Tennessee
  - SUN-131-03 Investigational Site, Nashville, Tennessee
  - SUN-131-03 Investigational Site, Cedar Park, Texas
  - SUN-131-03 Investigational Site, Houston, Texas
  - SUN-131-03 Investigational Site, Lakeway, Texas
  - SUN-131-03 Investigational Site, Mission, Texas
  - SUN-131-03 Investigational Site, San Antonio, Texas
  - SUN-131-03 Investigational Site, Salt Lake City, Utah
  - SUN-131-03 Investigational Site, Exmore, Virginia
  - SUN-131-03 Investigational Site, Falls Church, Virginia
  - SUN-131-03 Investigational Site, Norfolk, Virginia
  - SUN-131-03 Investigational Site, Racine, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo TDS: Placebo TDS was applied for a minimum of 16 hours and a maximum of 24 hours each day for 14 days.
- SUN-131 1.5% TDS: SUN-131 1.5% TDS was applied for a minimum of 16 hours and a maximum of 24 hours each day for 14 days.
Period: Overall Study
Arm/Group | Placebo TDS | SUN-131 1.5% TDS
Started | 131 | 132
Completed | 116 | 120
Not Completed | 15 | 12

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized subjects who received the study drug. Intent-to-treat (ITT) population included all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo TDS | SUN-131 1.5% TDS | Total
Number analyzed (Participants) | 131 | 132 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (17.00) | 49.0 (16.03) | 47.9 (16.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 81 | 163
  Male | 49 | 51 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 88 | 90 | 178
  Black or African American | 36 | 31 | 67
  Asian | 3 | 3 | 6
  American Indian or Alaskan Native | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Multi-racial (no primary race) | 1 | 3 | 4
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 131 | 132 | 263

OUTCOME MEASURES:

1. Primary Outcome: The Proportions of Participants Who Experienced Complete Response of the Study Chalazion by Day 15 ± 1
Description: Complete response was defined as the absence of any significant clinical signs of a chalazion, based on clinical judgment by an investigator.
Time Frame: Baseline to Day 15 ± 1
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo TDS | SUN-131 1.5% TDS
Number analyzed (Participants) | 131 | 132
Participants | 28 | 32
Statistical Analysis 1: Comparison: Placebo TDS vs SUN-131 1.5% TDS; Test type: Superiority; p = 0.579, 2-sided Pearson's chi-square

2. Secondary Outcome: The Proportions of Participants Who Experienced Complete Response of the Study Chalazion With Upper Eyelid by Day 15 ± 1
Description: as for outcome 1
Time Frame: Baseline to Day 15 ± 1
Population: Intent-to-treat (ITT) population included all randomized participants with upper eyelid chalazion.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo TDS | SUN-131 1.5% TDS
Number analyzed (Participants) | 81 | 95
Participants | 14 | 27
Statistical Analysis 1: Comparison: Placebo TDS vs SUN-131 1.5% TDS; Test type: Superiority; p = 0.082, 2-sided Pearson's chi-square

ADVERSE EVENTS:
Time Frame: The reporting period for AEs started after the first study drug application on Day 1 and ended at Follow-up Telephone Contact (Day 22 ± 3).
Description: A Treatment-Emergent Adverse Event (TEAE) is an adverse event with a start date on or after the initial dose of study drug and up to 5 days after the last dose of study drug.
Arm/Group | Placebo TDS | SUN-131 1.5% TDS
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/132
Other Adverse Events (participants affected / at risk) | 19/131 | 23/132
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo TDS (N=131) | SUN-131 1.5% TDS (N=132)
Chalazion (Eye disorders) | 4 (6) | 2 (2)
Conjunctival follicles (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Pinguecula (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eyelid disorder (Eye disorders) | 0 (0) | 1 (2)
Eyelid pain (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Application site discomfort (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator will not disclose information regarding this clinical investigation, or publish results of the investigation without authorization from Senju USA, Inc.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT03248440/Prot_SAP_000.pdf